CLINICAL TRIAL: NCT05346588
Title: Feasibility Study for the Trajectories of Recovery After Intravenous Propofol Versus Inhaled VolatilE Anesthesia (THRIVE) Trial
Brief Title: THRIVE Feasibility Trial
Acronym: THRIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Michigan (Other); University of Pennsylvania (Other); Stanford University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Michael Avidan, Prof of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 202205053
Record Dates: First submitted 2022-03-11; First posted 2022-04-26 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Surgery--Complications; Anesthesia Complication; Anesthesia Awareness; Anesthesia Emergence Delirium; Anesthesia; Surgery; Quality of Life; Pain, Postoperative; Nausea, Postoperative; Anesthesia Morbidity; Depression; Sleep Disorders, Circadian Rhythm
Keywords: Quality of recovery; Intraoperative awareness
MeSH Terms: conditions — Intraoperative Awareness; Emergence Delirium; Pain, Postoperative; Postoperative Nausea and Vomiting; Depression; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol total intravenous anesthesia (TIVA) (Active Comparator): No administration of inhaled agent.
  Interventions: Other: Anesthetic technique Propofol TIVA
- Inhaled volatile general anesthesia (Active Comparator): Must administer inhaled agent.
  Interventions: Other: Anesthetic technique inhaled agent

INTERVENTIONS:
Other: Anesthetic technique Propofol TIVA — Propofol TIVA no inhaled agent
  Other Names: Propofol TIVA
  Arms: Propofol total intravenous anesthesia (TIVA)
Other: Anesthetic technique inhaled agent — must administer inhaled agent.
  Other Names: Inhaled agent
  Arms: Inhaled volatile general anesthesia

SUMMARY:
To evaluate the feasibility of a pragmatic, large scale, comparative effectiveness, randomized evaluation of patient experience of intravenous propofol versus inhaled volatile anesthesia.

DETAILED DESCRIPTION:
Two-center single-blinded randomized feasibility study, with randomization 1:1 to either propofol TIVA or inhaled volatile general anesthesia for patients who are receiving elective non-cardiac surgery. Patients will be stratified by clinical site with 150 participants per site.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing elective non-cardiac surgery expected to last ≥ 60 min requiring general anesthesia, including a tracheal tube or laryngeal mask airway (or similar supra-glottic device)

Exclusion Criteria:

* Inability to provide informed consent in English
* Pregnancy (based on patient report or positive test on the day of surgery)
* Surgical procedure requiring general, regional, neuraxial anesthesia administered by an anesthesia clinician (anesthesiologist, CRNA, anesthesiology assistant) occurring within 30 days prior to or planned to occur within 30 days after surgery date
* Contraindication to propofol TIVA or inhaled volatile (for example, documented allergy to propofol, history of severe postoperative nausea or vomiting, concern for or history of malignant hyperthermia)
* Surgical procedures requiring specific general anesthesia option (for example, TIVA required for neuromonitoring).
* Hospital approved, written protocol mandating a particular technique
* History of intraoperative awareness during general anesthesia based on patient self-report on the day of consent
* Planned postoperative intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Proportion participating | 8 months
  Proportion of patients who are approached to participate by the study team and who consent to participate in the study.
Proportion receiving TIVA | 8 months
  Proportion of patients in the propofol TIVA group who receive per protocol treatment (i.e. they receive no inhaled agents as part of their anesthetic).
Proportion receiving inhaled anesthesia | 8 months
  Proportion of patients in the inhaled volatile group who receive per protocol treatment (i.e. they do receive inhaled agents as part of their anesthetic).

SECONDARY OUTCOMES:
Completeness of data collection | 11 months
  Completeness of data collection (defined as the percentage of instruments or data fields completed with at least 90% of expected forms or relevant fields completed at each time point and with each instrument)

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Kheterpal, MD, Principal Investigator — University of Michigan; Michael S Avidan, MBBcH, Principal Investigator — Washington Univeristy
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Hosptial of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tellor Pennington BR, Colquhoun DA, Neuman MD, Politi MC, Janda AM, Spino C, Thelen-Perry S, Wu Z, Kumar SS, Gregory SH, Avidan MS, Kheterpal S; THRIVE research group. Feasibility pilot trial for the Trajectories of Recovery after Intravenous propofol versus inhaled VolatilE anesthesia (THRIVE) pragmatic randomised controlled trial. BMJ Open. 2023 Apr 17;13(4):e070096. doi: 10.1136/bmjopen-2022-070096. PMID 37068889